CLINICAL TRIAL: NCT02876653
Title: Accelerated Aging in Middle-Aged Men With Sleep-disordered Breathing.
Acronym: SAOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: P091110
Record Dates: First submitted 2016-07-31; First posted 2016-08-24 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-07

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive sleep apnea; Aging; Telomere length
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Severe OSA (Other): Patients with severe OSA (AHI > 30)
  Interventions: Other: Polysomnography , blood collection, bone densitometry and Functional respiratory explorations
- Moderate OSA (Other): Patients with moderate OSA (5 < AHI ≤ 30)
  Interventions: Other: Polysomnography , blood collection, bone densitometry and Functional respiratory explorations
- Healthy volunteers (Other): Healthy volunteers (AHI ≤ 5)
  Interventions: Other: Polysomnography , blood collection, bone densitometry and Functional respiratory explorations

INTERVENTIONS:
Other: Polysomnography , blood collection, bone densitometry and Functional respiratory explorations — Blood collection, Bone densitometry and Functional respiratory explorations are a specific interventions of protocol for the 3 arms. Polysomnography is a specific intervention for the arms " healthy volunteers "

SUMMARY:
Obstructive Sleep Apnea Syndrome (OSAS) regardless of any other associated risk factor can lead to accelerated aging. The study of aging-related Obstructive Sleep Apnea (OSA) is difficult because of associated risk factors (diabetes, hypertension, dyslipidemia, obesity), promoting themselves aging. The investigators propose to compare a group of OSAS patients free of any associated pathology, to subjects matched for age, sex, smoking and body mass index (BMI)

ELIGIBILITY:
Inclusion Criteria

Patient:

* Men aged 20 to 65 years
* Having polysomnography in the Functional Explorations department, Sleep Laboratory, Hospital Henri Mondor, Creteil
* With an AHI > 5 / h

Healthy volunteers:

* Men aged 20 to 65 years
* With an AHI ≤ 5 / h

Exclusion Criteria

All subjects:

* Known cardiovascular risk: hypertension treated, diabetes treated, dyslipidemia treated,
* Known cardiovascular disease associated (heart failure, rhythm disorder ...)
* Known respiratory diseases
* Known neoplastic pathology, known chronic inflammatory disease
* Psychiatric pathology treated
* Medication
* Not affiliated to the French social health care system
* Major protected person
* Private person of liberty
* People in emergency situation
* Patient refusing to participate in the study

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2011-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Telomere length of circulating leukocytes | 4 weeks

SECONDARY OUTCOMES:
Carotid-femoral pulse wave velocity | 4 weeks
Bone density | 4 weeks
Correlation between biological parameters and neuropsychological assessment | 4 weeks
Markers of oxidative stress: Malondialdehyde, heme oxygenase-1 | 4 weeks
Markers of inflammation: hs-CRP, IL-6, IL-8, MCP-1 | 4 weeks
Markers of growth hormone axis (GH, IGF-1, IGFBP) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Boyer, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France